CLINICAL TRIAL: NCT04672629
Title: Clinical Profile of Neonates Diagnosed by Echocardiography as Having Patent Ductus Arteriousus in Assiut University Hospital for Children
Brief Title: Clinical Profile of Neonates Having Patent Ductus Arteriosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Emad Amin, doctor, Assiut University
Other Study IDs: PDA in neonatology
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2020-12

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: echocardiography — follow up echocardiography

SUMMARY:
The study aims to evaluate the clinical presentation and course of PDA diagnosed at neonatal period in the neonatology unit of Assiut University Hospital for Children.

DETAILED DESCRIPTION:
One of the most common cardiovascular problems that prematurely born infants experience early in life is patent ductus arteriosus (PDA).

The ductus arteriosus is a blood vessel that connects the two major arteries, namely the aorta and the pulmonary artery, and is essential in maintaining circulation in fetal life. After the baby is born and the fetal circulation changes to adult circulation, the ductus arteriosus functionally closes between 18 and 24 hours of life (1 ).

The arterial duct is a fetal blood vessel that is programmed to close shortly after birth. If the vessel remains patent beyond 3 months of life (a persistently patent arterial duct) it can result in volume loading of the left heart and should be closed either surgically or by a catheter-based procedure. A patent arterial duct is common in the newborn, particularly premature infants, and can contribute to persistent respiratory problems. (2) Historical estimates have placed the incidence of isolated PDA at approximately 0.05% of all live births. Isolated PDA accounts for 5% to 10% of congenital heart defects (3) number most likely represents the prevalence of a "symptomatic" PDA-that is, one that results in evidence of increased pulmonary blood flow, left heart volume overload, elevated PA pressure, murmur, etc. With the advent of color Doppler echocardiography, the incidental recognition of asymptomatic "silent" ductus has become more common. Some have estimated the prevalence of silent PDA among children and adults to be up to 0.5%, far more common than the "symptomatic" PDA (4).

However, in babies born prematurely, the ductus arteriosus often fails to close spontaneously and leads to a number of morbidities. it has been shown that in infants born with a birth weight of <1000 g, the ductus arteriosus remains open in 66% of infants beyond the ﬁrst week of life. In the extreme premature population born at 24 weeks of gestation, only 13% of infants are found to have their ductus closed by the end of the ﬁrst week (5).This makes PDA an important issue from the clinical management perspective in the ﬁrst few days of life in preterm infants.

It is associated with a number of comorbidities such as necrotising enterocolitis (NEC), bronchopulmonary dysplasia and intraventricular haemorrhage (IVH) (6-7).

The management controversy has mainly focused on when to treat and with what to treat. To increase the complexity of m atters, these two aspects of PDA management are not mutually exclusive, with the modality of treatment often being dictated by the timing of treatment. There have been a large number of published studies, meta-analyses and editorials focusing on different aspects of management.(8-9)Regarding the timing of treatment, prophylactic therapy has gradually fallen out of favor and neonatal units have shifted towards a more conservative approach by treating only the clinically and echocardiographically (ECHO) signiﬁcant PDA (10).However, the big dilemma that still persists among neonatologists is what to use as the primary modality of treatment.

ELIGIBILITY:
Inclusion Criteria:

- 1- Neonatal period (0-28 days) including fullterm and preterm infants for whom echocardiography is indicated.

2- Absence of other congenital cardiac defects.

Exclusion Criteria:

* PDA associated with other cardiac anomalies.

Ages: 0 Days to 28 Days | Sex: All
Age Groups: Child
Study Population: 1- Neonatal period (0-28 days) including fullterm and preterm infants for whom echocardiography is indicated
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Determine the percentage of cases with PDA admitted to our neonatology unit per year. | one year
  This study was proposed to improve practice in our neonatal unit regarding interpretation of echocardiograms showing the diagnosis of PDA and decisions based on.

REFERENCES:
- [Background] Vettukattil JJ. Pathophysiology of Patent Ductus Arteriosus in the Preterm Infant. Curr Pediatr Rev. 2016;12(2):120-2. doi: 10.2174/157339631202160506002215. PMID 27197953
- [Background] Louis D, ElSayed YN, Ojah C, Alvaro R, Shah PS, Dunn M; Canadian Neonatal Network Investigators. Predictors of PDA Treatment in Preterm Neonates Who Had Received Prophylactic Indomethacin. Am J Perinatol. 2018 Apr;35(5):509-514. doi: 10.1055/s-0037-1608792. Epub 2017 Nov 28. PMID 29183097